CLINICAL TRIAL: NCT04012450
Title: The Effects of Combined Spinal-epidural Anesthetics During Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, SAAR AHARONI MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0500-15-RMB
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural Anesthesia (Active Comparator): Women in labor receiving epidural anesthesia
  Interventions: Procedure: Epidural anesthesia
- Spinal-epidural (Active Comparator): Women in labor receiving spinal-epidural anesthesia
  Interventions: Procedure: spina-epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — Performing an epidural anesthesia
  Arms: Epidural Anesthesia
Procedure: spina-epidural anesthesia — Performing a spina-epidural anesthesia
  Arms: Spinal-epidural

SUMMARY:
Women who fulfil the inclusion criteria and who intended to regional anesthesia will be randomized into the epidural anesthesia arm or to the spinal-epidural anesthesia arm. Sonographic evaluation of the flow in the uterine artery, umbilical artery, and middle cerebral artery will be documented to each patient prior and following the regional anesthesia.

DETAILED DESCRIPTION:
Patients will receive information regarding the available anesthesia during labor that are available in the delivery room including regional and systemic.

After receiving the patient informed consent for regional anesthesia (epidural or spinal-epidural), patients will be offered to participate in our study.

After receiving the patients' informed consent for participating in the study, patients will be randomized to either the epidural anesthesia group or to the spinal-epidural anesthesia group.

A doppler ultrasound will be performed on each patient prior to and following the regional anesthesia, the flow in the uterine artery, umbilical artery, and the middle cerebral artery of the fetus will be recorded.

Demographic and obstetrical information will be collected from the patients' electronic files.

ELIGIBILITY:
Inclusion criteria:

Gestational age of 37 and above Singleton Vertex presentation Desired regional anesthesia

Exclusion criteria:

Contraindication to regional anesthesia Placental abnormalities (placenta previa, placenta accreta, placental separation) Pregnancy following fetal reduction or intrauterine fetal death (IUFD) Fetal malformations Intrauterine growth retardation (IUGR) Suspected chorioamnionitis (including body temperature above 38.5 degrees Celsius)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Uterine artery flow | Up to 48 hours from onset of anesthesia
  Changes in uterine artery flow before and after regional anesthesia
Umbilical artery flow | Up to 48 hours from onset of anesthesia
  Changes in umbilical artery flow before and after regional anesthesia
Middle cerebral artery flow | Up to 48 hours from onset of anesthesia
  Changes in middle cerebral artery flow before and after regional anesthesia

SECONDARY OUTCOMES:
Fetal heart rate abnormalities | Up to 48 hours from onset of anesthesia
  Fetal heart rate deceleration
Fetal bradycardia within 1 hour | Up to one hour from onset of anesthesia
  Fetal bradycardia
Mode of delivery | Up to delivery
  Mode of delivery - vaginal/instrumental/cesarean section
Meconial amniotic fluid | Up to delivery
  Meconial amniotic fluid
Umbilical artery blood acidity level (PH) | Immediate after delivery
  Umbilical artery blood PH
Apgar at 1 and 5 minutes | Up to 5 minutes from delivery
  Apgar at 1 and 5 minutes
Admission to Neonatal Intensive Care Unit (NICU) | Up to 72 hours from delivery
  Admission to NICU

CONTACTS AND LOCATIONS:
Overall Officials: Saar Aharoni, MD, Principal Investigator — Rambam Heath-Care Campus

IPD SHARING:
Plan to Share IPD: Undecided